CLINICAL TRIAL: NCT04276233
Title: A Phase 4, Open-label, Single Arm, 24-week, Study to Evaluate the Safety and Efficacy of Mepolizumab 100 mg SC Administered Every 4 Weeks in Indian Participants Aged ≥18 Years With Severe Eosinophilic asthMa (PRISM)
Brief Title: Efficacy and Safety Study of Mepolizumab 100 Milligram (mg) Subcutaneous (SC) in Indian Participants Aged Greater Than or Equal to (>=) 18 Years With Severe Eosinophilic Asthma
Acronym: PRISM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Tech Observer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209682
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Asthma
Keywords: Mepolizumab; Oral corticosteroids; Prednisolone; Prednisone; Severe Eosinophilic asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab; Albuterol

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with severe eosinophilic asthma (Experimental): Participants with severe eosinophilic asthma will receive Mepolizumab 100 mg subcutaneously into the upper arm or thigh every 4 weeks for a period of 24 weeks (total of 6 doses). Salbutamol metered dose inhalers (MDIs) will be provided as rescue medication during treatment period.
  Interventions: Drug: Mepolizumab; Drug: Salbutamol

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab will be available as a lyophilized cake in sterile vials and will be reconstituted with sterile water for injection, just prior to use.
Drug: Salbutamol — Salbutamol metered dose inhalers (MDIs) will be provided as rescue medication during treatment period.

SUMMARY:
Mepolizumab is a humanized monoclonal antibody (IgG1, kappa) that blocks interleukin- 5 (IL-5) thus inhibits production and survival of eosinophils. The aim of this phase 4, open-label, single-arm study is to evaluate the safety and efficacy of Mepolizumab 100 mg SC administered every 4 weeks in Indian participants aged 18 years or above with severe eosinophilic asthma. After the first dose of mepolizumab, participants will receive 5 more doses of mepolizumab at 4 weekly intervals. Following the last dose of mepolizumab, the end of the study Visit will occur 4 weeks later. During the treatment period, OCS use and dose adjustment in participants will be as per the investigator's discretion and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to (≥) 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Asthma: Evidence of asthma as documented by either: (a) Airway reversibility (FEV1>=12% and 200 milliliter (ml) demonstrated at Visit 1 (screening) or Visit 2 (Week 0) OR documented in the previous 12 months OR (b) Airway hyperresponsiveness (methacholine: PC20 of <8mg/mL or histamine: PD20 of <7.8 μmol; mannitol: decrease in FEV1 as per the labelled product instructions) documented in the 12 months prior to Visit 2 (Week 0) OR (c) Airflow variability in clinic FEV1 >=20% between two consecutive clinic visits documented in the 12 months prior to Visit 2 (FEV1 recorded during an exacerbation should not be considered for this criteria) OR (d) Airflow variability as indicated by >20% diurnal variability in peak flow observed on 3 or more days during the optimization period.
* Participants with Eosinophilic asthma: prior documentation of eosinophilic asthma or high likelihood of eosinophilic asthma as FEV1: Persistent airflow obstruction as indicated by: For participants >=18 years of age at Visit 1 (screening) or Visit 2 (Week 0), a pre- bronchodilator FEV1 <80% predicted. For predicted FEV1 values National Health and Nutrition Examination Survey (NHANES) III values will be used and adjustments to these values will be made for race.
* Eosinophilic Phenotype: Airway inflammation characterized as eosinophilic in nature as indicated by one of the following characteristics: (a) An elevated peripheral blood eosinophil level of >=300 cells/microliter(μL) that is related to asthma within the previous 12 months prior to Visit 2 (Week 0). OR (b) Peripheral baseline eosinophil level >=150 cells/μL between Visit 1 (screening) and Visit 2 (Week 0) that is related to asthma.
* Participants eligible for mepolizumab treatment as per independent clinical judgment of treating physician in alignment with local prescribing information.
* Inhaled Corticosteroids: requirement for regular treatment with high dose inhaled corticosteroid in the 6 months prior to Visit 1 (screening). For 18 years of age and older: Inhaled corticosteroids (ICS) dose must be >=880 microgram (mcg)/day fluticasone propionate (FP) (ex-actuator) or equivalent daily.
* Controller Medication: Current treatment with an additional controller medication for at least 3 months OR having used and failed an additional controller medication for at least 3 successive months during the prior 12 months [e.g., long-acting beta2-agonist (LABA), leukotriene receptor antagonist (LTRA), or theophylline].
* Male or eligible female. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: (a) Is not a woman of childbearing potential (WOCBP) OR (b) Is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1% during the intervention period and for at least 16 weeks after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. (c) A WOCBP must have a negative highly sensitive pregnancy test (serum) within 8 weeks before the first dose of study intervention. (d) Additional requirements for pregnancy testing during and after study intervention are located. (e) The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Treatment Period Criteria

* Eosinophilic asthma: Prior documentation of eosinophilic asthma or high likelihood of eosinophilic asthma.
* eDiary Compliance: Compliance with completion of the eDiary defined as: (a) Completion of symptom scores on 4 or more days out of the last 7 days immediately preceding Visit 2 (Week 0). (b) Completion of information relating to rescue medication use on 4 or more days out of the last 7 days immediately preceding Visit 2 (Week 0). (c) Completion of PEF measurements on 4 or more days out of the last 7 days immediately preceding Visit 2 (Week 0).

Exclusion Criteria:

* Concurrent Respiratory Disease: Presence of a clinically important lung condition other than asthma. This includes but is not limited to current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior screening (Participants who had localized carcinoma (i.e. basal or squamous cell) of the skin which was resected for cure will not be excluded).
* Liver Disease: Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, and known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Cardiovascular: Participants who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment. Including but not limited to: (a) known ejection fraction of <30% OR (b) severe heart failure meeting New York Heart Association Class IV OR (c) hospitalized in the 12 months prior to Visit 1 (screening) for severe heart failure meeting New York Heart Association Class III OR (d) angina diagnosed less than 3 months prior to Visit 1 (screening) or at Visit 1.
* Other Concurrent Medical Conditions: Participants who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
* Eosinophilic Diseases: Participants with other conditions that could lead to elevated eosinophils such as Hypereosinophilic Syndromes, including Churg-Strauss Syndrome, or Eosinophilic Esophaghitis. Participants with a known, pre-existing parasitic infestation within 6 months prior to Visit 1 (screening) are also to be excluded.
* Omalizumab Use: Participants who have received omalizumab within 130 days of Visit 1 (screening).
* Other Monoclonal Antibodies: Participants who have received any monoclonal antibody (other than omalizumab) to treat inflammatory disease within 5 half-lives of Visit 1 (screening).
* Investigational Medications: Participants who have received treatment with an investigational drug within the past 30 days or five terminal phase half-lives of the drug whichever is longer, prior to Visit 1 (this also includes investigational formulations of marketed products).
* Participants who have previously participated in any study of mepolizumab and received Investigational Product (including placebo).
* ECG: ECG assessment QTcF > 450msec or QTcF > 480 msec for participants with Bundle Branch Block. Participants are excluded if an abnormal ECG finding from the 12-lead ECG conducted at Screening (Visit 1) is considered to be clinically significant and would impact the participant's participation during the study, based on the evaluation of the Investigator.
* Immunodeficiency: A known immunodeficiency (e.g. human immunodeficiency virus - HIV), other than that explained by the use of corticosteroids taken as therapy for asthma.
* Smoking history: Current smokers or former smokers with a smoking history of >=10 pack years. A former smoker is defined as a participant who quit smoking at least 6 months prior to Visit 1 (screening).
* Hypersensitivity: Participants with a known allergy or intolerance to a monoclonal antibody or biologic.
* Pregnancy: Participants who are pregnant or breastfeeding. Patients should not be enrolled if they plan to become pregnant during the time of study participation.
* Alcohol/Substance Abuse: A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1 (screening).
* Adherence: Participants who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.

Treatment Period Criteria

* Laboratory abnormality: Evidence of clinically significant abnormality in the haematological, biochemical or urinalysis screen at Visit 1 (screening), as judged by the investigator.
* Alanine transferase (ALT) >2 x upper limit of normal (ULN).
* Bilirubin > 1.5 x ULN (isolated bilirubin>1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* No cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice. Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B or C e.g., presence of hepatitis B surface antigen [HBsAg] or positive hepatitis C antibody test result) is acceptable if the participant otherwise meets eligibility criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- India (10):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Byculla Mumbai
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Kanpur
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Noida
  - GSK Investigational Site, Pune

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the safety and efficacy of Mepolizumab in participants with severe eosinophilic asthma.
Pre-assignment Details: A total of 100 participants were enrolled in the study.
Groups:
- Mepolizumab 100 mg SC: Participants with severe eosinophilic asthma received mepolizumab 100 milligrams (mg) subcutaneously (SC) into the upper arm, thigh or abdomen every 4 weeks for a period of 24 weeks (total of 6 doses). Salbutamol metered dose inhalers (MDIs) were provided as a rescue medication during treatment period.
Period: Overall Study
Arm/Group | Mepolizumab 100 mg SC
Started | 100
Completed | 90
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Any untoward medical occurrence that, at any dose that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment was categorized as SAE. Adverse events which were not serious were considered as non-serious adverse events. Number of participants with SAEs and common (greater than equal to [>=] 3 percent [%]) non-SAEs were reported.
Time Frame: Up to Week 24
Population: Safety Population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 100
Participants
  SAEs | 3
  Non-SAEs | 9

2. Secondary Outcome: Number of Participants With Clinically Significant Exacerbations (Including Exacerbations Requiring Hospitalization or Emergency Department [ED Visits])
Description: Clinically significant exacerbations of asthma were defined as worsening of asthma which requires use of systemic corticosteroids and/or hospitalization and/or ED visits. Exacerbations were treated per the investigator's clinical practice protocol with the use of oral or parenteral corticosteroids. Clinically significant exacerbations were recorded in the electronic case report form (eCRF) by the Investigator or designee were verified using data from the electronic Diary. Number of participants with clinically significant exacerbations were reported.
Time Frame: Up to Week 24
Population: Safety Population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 100
Participants | 8

3. Secondary Outcome: Number of Participants With Exacerbations Requiring Hospitalization or ED Visits
Description: Exacerbations of asthma are defined as worsening of asthma which requires use of systemic corticosteroids and/or hospitalization and/or ED visits. Number of participants with exacerbations requiring hospitalization or ED visits were reported.
Time Frame: Up to Week 24
Population: Safety Population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 100
Participants | 2

4. Secondary Outcome: Number of Participants With Exacerbations Requiring Hospitalization
Description: Exacerbations of asthma are defined as worsening of asthma which requires use of systemic corticosteroids and/or hospitalization. Number of participants with exacerbations requiring hospitalization were reported.
Time Frame: Up to Week 24
Population: Safety Population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 100
Participants | 2

5. Secondary Outcome: Change From Baseline in Clinic Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Week 24
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 was measured electronically by spirometry. Baseline is defined as the value recorded at pre-dose (Weeks -2 to -1) assessment. The change from Baseline in pre-bronchodilator FEV1 was calculated as the value at Week 24 minus the value at Baseline.
Time Frame: Baseline (Weeks -2 to -1) and Week 24
Population: Safety Population included all participants who took at least 1 dose of study intervention. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 86
Liters | 0.081 (0.0667)

6. Secondary Outcome: Change From Baseline in Clinic Post-bronchodilator FEV1 at Week 24
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 was measured electronically by spirometry. Baseline is defined as the value recorded at pre-dose (Weeks -2 to -1) assessment. The change from Baseline in post-bronchodilator FEV1 was calculated as the value at Week 24 minus the value at Baseline.
Time Frame: Baseline (Weeks -2 to -1) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 83
Liters | 0.055 (0.0555)

7. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score at Week 24
Description: The ACQ-5 is a five-item questionnaire, designed to be self-completed by the participants. The five questions (nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms. The response options for all these questions consists of a zero (no impairment/limitation) to six (total impairment/ limitation). The ACQ-5 score is calculated as the mean of these 5 item responses and ranges from scores 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicate lower asthma control. Baseline is defined as the value recorded at pre-dose (Weeks -2 to -1) assessment. The change from Baseline was calculated as the value at Week 24 minus the Baseline value.
Time Frame: Baseline (Weeks -2 to -1) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 86
Scores on a scale | -0.69 (0.121)

8. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (PEF) During Weeks 21 to 24
Description: PEF was defined as the maximum speed of expiration of a participant, measured with electronic peak flow meter. Baseline is defined as the value recorded at pre-dose (Weeks -2 to -1) assessment. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Weeks -2 to -1) and Weeks 21 to 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters per minute (L/min)
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 85
Liters per minute (L/min) | 13.67 (5.330)

9. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs were adverse events associated with the identified and potential risks of mepolizumab. AESIs were systemic/ local site reactions, all infections (Infections from Infections and infestations System Organ Class [SOC]), opportunistic infections, neoplasm, malignancies, cardiac disorders and serious cardiac, vascular and thromboembolic (CVT) events.
Time Frame: Up to Week 24
Population: Safety Population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 100
Participants
  Systemic/local site reactions | 3
  All infections | 5
  Opportunistic infections | 0
  Neoplasm | 0
  Malignancies | 0
  Cardiac disorders | 0
  Serious cardiac, vascular and thromboembolic (CVT) events | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and common (>=3%) non-serious adverse events (non-SAEs) were collected up to Week 24
Description: All-cause mortality, SAEs and non-SAEs were reported for the Safety Population which included all participants who took at least 1 dose of study intervention.
Arm/Group | Mepolizumab 100 mg SC
All-Cause Mortality (participants affected / at risk) | 1/100
Serious Adverse Events (participants affected / at risk) | 3/100
Other Adverse Events (participants affected / at risk) | 9/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 100 mg SC (N=100)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 100 mg SC (N=100)
Pyrexia (General disorders) | 5
Headache (Nervous system disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT04276233/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04276233/SAP_001.pdf